CLINICAL TRIAL: NCT03151486
Title: A Double-Blind, Placebo-Controlled, Randomized Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-55308942 in Healthy Male and Female Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-55308942 in Healthy Male and Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108293; 2017-000303-25 (EudraCT Number); 55308942EDI1001 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2017-04-26; First posted 2017-05-12 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-55308942

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1:JNJ-55308942 0.5 mg or Placebo (SAD Part) (Experimental): Participants will be randomized to receive a single dose of JNJ-55308942 0.5 milligrams (mg) or matching placebo as an oral solution after an overnight fast on Day 1 of Cohort 1 after single ascending dose (SAD).
  Interventions: Drug: JNJ-55308942 0.5 mg; Drug: Placebo
- Cohort 2: JNJ-55308942 1.5 mg or Placebo (SAD Part) (Experimental): Participants will be randomized to receive a single dose of JNJ-55308942 1.5 mg or matching placebo as an oral solution after an overnight fast on Day 1.
  Interventions: Drug: JNJ-55308942 1.5 mg; Drug: Placebo
- Cohort 3: JNJ-55308942 4 mg or Placebo (SAD Part) (Experimental): Participants will be randomized to receive a single dose of JNJ-55308942 4 mg or matching placebo as an oral solution after an overnight fast on Day 1.
  Interventions: Drug: JNJ-55308942 4 mg; Drug: Placebo
- Cohort 4: (JNJ-55308942 12 mg or Placebo (SAD Part)) (Experimental): Participants will be randomized to receive a single dose of JNJ-55308942 12 mg or matching placebo as an oral solution after an overnight fast on Day 1.
  Interventions: Drug: JNJ-55308942 12 mg; Drug: Placebo
- Cohort 5: JNJ-55308942 36 mg or Placebo (SAD Part) (Experimental): Participants will be randomized to receive a single dose of JNJ-55308942 36 mg or matching placebo as an oral solution after an overnight fast on Day 1.
  Interventions: Drug: JNJ-55308942 36 mg; Drug: Placebo
- Cohort 6: JNJ-55308942 100 mg or Placebo (SAD Part) (Experimental): Participants will be randomized to receive a single dose of JNJ-55308942 100 mg or matching placebo as an oral solution after an overnight fast on Day 1.
  Interventions: Drug: JNJ-55308942 100 mg; Drug: Placebo
- Cohort 7: JNJ-55308942 or Placebo (SAD Part) (Experimental): Participants will be randomized to receive a single dose of JNJ-55308942 or matching placebo as an oral solution in a fed state on Day 1. The dose selected for this cohort will be based on the data obtained from the single ascending dose cohorts.
  Interventions: Drug: JNJ-55308942: Fed State; Drug: Placebo
- Cohort 1: JNJ-55308942 or Placebo (MAD Part) (Experimental): Participants will be randomized to receive JNJ-55308942 or matching placebo once daily as an oral solution for 10 consecutive days (Day 1 to 10). The doses for the multiple ascending doses (MAD) will be determined based on the data from the SAD part.
  Interventions: Drug: JNJ-55308942: MAD Part; Drug: Placebo
- Cohort 2: JNJ-55308942 or Placebo (MAD Part) (Experimental): Participants will be randomized to receive JNJ-55308942 or matching placebo once daily as an oral solution for 10 consecutive days (Day 1 to 10). The doses for the MAD will be determined based on the data from the SAD part.
  Interventions: Drug: JNJ-55308942: MAD Part; Drug: Placebo
- Cohort 3: JNJ-55308942 or Placebo (MAD Part) (Experimental): Participants will be randomized to receive JNJ-55308942 or matching placebo once daily as an oral solution for 10 consecutive days (Day 1 to 10). The doses for the MAD will be determined based on the data from the SAD part.
  Interventions: Drug: JNJ-55308942: MAD Part; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-55308942 0.5 mg — Participants will receive JNJ-55308942 0.5 mg as an oral solution after an overnight fast on Day 1.
  Arms: Cohort 1:JNJ-55308942 0.5 mg or Placebo (SAD Part)
Drug: JNJ-55308942 1.5 mg — Participants will receive JNJ-55308942 1.5 mg as an oral solution after an overnight fast on Day 1.
  Arms: Cohort 2: JNJ-55308942 1.5 mg or Placebo (SAD Part)
Drug: JNJ-55308942 4 mg — Participants will receive JNJ-55308942 4 mg as an oral solution after an overnight fast on Day 1.
  Arms: Cohort 3: JNJ-55308942 4 mg or Placebo (SAD Part)
Drug: JNJ-55308942 12 mg — Participants will receive JNJ-55308942 12 mg as an oral solution after an overnight fast on Day 1.
  Arms: Cohort 4: (JNJ-55308942 12 mg or Placebo (SAD Part))
Drug: JNJ-55308942 36 mg — Participants will receive JNJ-55308942 36 mg as an oral solution after an overnight fast on Day 1.
  Arms: Cohort 5: JNJ-55308942 36 mg or Placebo (SAD Part)
Drug: JNJ-55308942 100 mg — Participants will receive a single oral dose of JNJ-55308942 100 mg as an oral solution after an overnight fast on Day 1.
  Arms: Cohort 6: JNJ-55308942 100 mg or Placebo (SAD Part)
Drug: JNJ-55308942: Fed State — Participants will receive JNJ-55308942 as an oral solution in fed state on Day 1. The dose selected for this cohort will be based on the data obtained from the single ascending dose cohorts.
  Arms: Cohort 7: JNJ-55308942 or Placebo (SAD Part)
Drug: JNJ-55308942: MAD Part — Participants will receive JNJ-55308942 once daily as an oral solution for 10 consecutive days (Day 1 to 10). The doses for the MAD will be determined based on the data from the SAD part.
  Arms: Cohort 1: JNJ-55308942 or Placebo (MAD Part); Cohort 2: JNJ-55308942 or Placebo (MAD Part); Cohort 3: JNJ-55308942 or Placebo (MAD Part)
Drug: Placebo — Participants will receive matching placebo in all cohorts.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics (PK) of JNJ-55308942 in healthy participants after administration of single and multiple oral doses.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m^2) (BMI = weight [kg] / height [m]^2), and a body weight of not less than 50 kilogram (kg)
* Participant must be healthy on the basis of physical examination, neurological examination, medical history, vital signs, and 12 lead (electrocardiogram) ECG, and peripheral capillary oxygen saturation [(SpO2) greater than or equal to (>=) 97 percent] performed at Screening and Day -1
* Participant must be healthy on the basis of clinical laboratory tests performed at Screening and Day -1. If the results of the serum chemistry panel, coagulation, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Female participants must not be of childbearing potential by fulfilling 1 of the criteria: a) be over 45 years of age with no menses for 12 months without an alternative medical cause, with screening follicle stimulating hormone (FSH) levels of greater than (>) 40 International Unit per Liter (IU/L) or milli-International Unit per milliliter (mIU/mL). b) be permanently surgically sterile. Permanent surgical sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy. Documentation of FSH levels is not required in the case of surgical sterility
* Female participants must have a negative serum pregnancy (Beta -human chorionic gonadotropin [Beta -hCG]) test at screening and a negative urine pregnancy test on Day -1

Exclusion Criteria:

* Participant has current, or history of, clinically significant medical illness including, but not limited to, liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Participant has a history of abnormal bleeding or clotting, or disorder of fibrinogen (example, dysfibrinogenemia, hypofibrinogenemia)
* Participant has history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the Investigator, with concurrence with the Sponsor's medical monitor, is considered cured with minimal risk of recurrence)
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 1 month or within a period of less than 10 times the drug's half-life, whichever is longer, before the planned first dose of study drug, or is currently enrolled in another investigational study
* Participant has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 5 years before Screening or positive test result(s) for alcohol or drugs of abuse (including barbiturates, opiates, cocaine, cannabinoids, amphetamines, ecstasy, phencyclidine, tricyclic antidepressants, and benzodiazepines) at Screening

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 6 Weeks
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Single Ascending Dose (SAD): Maximum Observed Plasma Concentration (Cmax) of JNJ-55308942 | Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours postdose on Day 1
  The Cmax is the maximum observed plasma concentration of JNJ-55308942.
SAD: Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-55308942 | Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours postdose on Day 1
  Tmax is defined as time to reach the maximum observed plasma JNJ-55308942 concentration.
SAD: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours Postdose (AUC [0-24]) of JNJ-55308942 | Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours postdose on Day 1
  AUC (0-24h) is defined as area under the plasma JNJ-55308942 concentration-time curve from time 0 to 24 hours postdose.
SAD: Area Under the Plasma Concentration-time Curve From Time Zero to Time of the Last Observed Quantifiable Concentration (AUC [0-Last]) of JNJ-55308942 | Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours postdose on Day 1
  AUC (0-last) is defined as area under the plasma JNJ-53308942 concentration-time curve from time 0 to time of the last observed quantifiable concentration.
SAD: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-55308942 | Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours postdose on Day 1
  AUC (0-infinity) is defined as area under the plasma JNJ-55308942 concentration-time curve from time 0 to infinite time.
SAD: Area Under the Plasma JNJ-55308942 Concentration-time Curve During a Dosing Interval (t) at steady-state (AUC tau) | Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours postdose on Day 1
  AUC tau is defined as area under the plasma JNJ-55308942 concentration-time curve during a dosing interval (tau) at steady-state.
SAD: Apparent elimination Half-Life (t1/2) of JNJ-55308942 | Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours postdose on Day 1
  The elimination half-life (T1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Multiple Ascending Dose (MAD): Maximum Observed Plasma Concentration (Cmax) of JNJ-55308942 on Day 1 | Predose, 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 16 hours postdose on Day 1
  The Cmax is the maximum observed plasma concentration of JNJ-55308942.
MAD: Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-55308942 on Day 1 | Predose, 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 16 hours postdose on Day 1
  Tmax is defined as time to reach the maximum observed plasma JNJ-55308942 concentration.
MAD: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours Postdose (AUC [0-24]) of JNJ-55308942 on Day 1 | Predose, 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 and 24 hours postdose on Day 1
  AUC (0-24h) is defined as area under the plasma JNJ-55308942 concentration-time curve from time 0 to 24 hours postdose.
MAD: Apparent elimination Half-Life (t1/2) of JNJ-55308942 on Day 1 | Predose, 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 16 hours postdose on Day 1
  The elimination half-life (T1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
MAD: Maximum Observed Plasma Concentration (Cmax) of JNJ-55308942 After Dosing on Day 10 | Predose, 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 and 120 hours postdose on Day 10
  The Cmax is the maximum observed plasma concentration of JNJ-55308942.
MAD: Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-55308942 After Dosing on Day 10 | Predose, 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 and 120 hours postdose on Day 10
  Tmax is defined as time to reach the maximum observed plasma JNJ-55308942 concentration.
MAD: Area Under the Plasma JNJ-55308942 Concentration-time Curve During a Dosing Interval (t) at steady-state (AUC tau) After Dosing on Day 10 | Predose, 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 and 120 hours postdose on Day 10
  AUC tau is defined as area under the plasma JNJ-55308942 concentration-time curve during a dosing interval (tau) at steady-state.
MAD: Apparent Elimination Half-Life (t1/2) of JNJ-55308942 After Dosing on Day 10 | Predose, 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96 and 120 hours postdose on Day 10
  The elimination half-life (T1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium